CLINICAL TRIAL: NCT02654106
Title: Fractionated Stereotactic Radiotherapy Combined With Temozolomide for Refractory Brain Metastases: A Single-arm, Single-center Phase II Trial
Brief Title: Stereotactic Radiotherapy Plus Temozolomide for Refractory Brain Metastases
Acronym: SRTRBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Cancer Foundation, China (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Dr, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-H&N-003
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Brain Metastases
Keywords: multiple brain metastases; large brain metastases; meningeal metastases; fractionated stereotactic radiotherapy; temozolomide
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refractory Brain Metastases (Experimental): Group A: multiple brain metastases: no less than 3 lesions in the brain Group B: Large Brain Metastases: the volume of lesion is no smaller than 6cc or the maximum diameter of the lesion is no shorter than 3cm Group C:Meningeal Metastases
  Interventions: Radiation: Fractionated Stereotactic Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: Fractionated Stereotactic Radiotherapy — The regular fraction modes were as follows: a. lesions≥3 cm：52Gy/4Gy/13f or 52.5Gy/3.5Gy/15f; b. lesions<2cm：36Gy/12Gy/3f or 24Gy/24Gy/1f; for lesions located in function areas, it would be adjusted to 40Gy/8Gy/5f; c. lesions 2-3cm：40-48Gy/8-10Gy/6-4f; d. lesions located in brainstem：50-60Gy/2.5-3Gy/20f.
  Other Names: FSRT
Drug: Temozolomide — concomitant TMZ: 75mg/m2 adjuvant TMZ: 150mg/m2*5d, q28d, 6cycles
  Other Names: TMZ

SUMMARY:
This clinical trial was designed to investigate the efficiency and toxicity of fractionated stereotactic radiotherapy(FSRT) combined with Temozolomide(TMZ) for refractory brain metastases.

DETAILED DESCRIPTION:
This is a single-arm, single center, phase II trial to investigate the feasibility and toxicity of FSRT plus TMZ for refractory brain metastases, which are defined as A: multiple brain metastases(≥3 lesions); B: large brain metastases(with one lesion's volume is no smaller than 6cc or the longest diameter is no shorter than 3cm); C: meningeal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of primary tumor and conformed brain metastases by enhanced MRI or CT
* the lesion number is no less than 3; or the tumor volume is no smaller than 6cc; or tumor diameter is no shorter than 3cm; or uncontrolled brain tumor after whole brain radiotherapy(WBRT); or the tumor is adjacent to essential structures of the brain, such as brain stem, optic chiasma, optic tract, etc.
* KPS ≥60，or KPS ≥40 and the limitation of motion is simply caused by brain tumor that is adjacent to the motor function areas.
* Age: 18-75 years old.
* Adequate end-organ function:

WBC≥4.0x109/L Neu ≥ 1.5x109/L Hemoglobin ≥ 110 g/L Platelets ≥100 x109/L Total bilirubin ≤ 1.5x ULN AST and ALT ≤ 1.5x ULN BUN and Cr: within the normal range

Exclusion Criteria:

* Other clinically significant diseases (e.g.myocardial infarction within the past 6 months, severe arrhythmia).
* Unable or unwilling to comply with the study protocol.
* The expected survival time is less than 3 months.
* Patients who are anticipated in other clinical trials of brain metastases.
* Patients who has been treated with SRT in other hospitals
* Pregnant patients or female patients whose HCG is positive
* Unsuitable to participate in study, that in the opinion of the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
intracranial progress free survival rate | up to 2 years
  defined as no progress of the treated lesions and no distant progress in the brain

SECONDARY OUTCOMES:
Overall survival rate | up to 3 year
progress free survival rate | up to 1 year
local control rate | up to 1 year
disease control rate (DCR) | 2-3 months after radiation
  Using RTOG9508 criteria, Tumor control is defined as CR+PR+SD
adverse event | from the day of radiation to the end of adjuvant TMZ，up to 6 months
  assessed by CTCAE criteria, v4.0 and RTOG criteria of the central nervous system
causes of death | from the day of radiation to death date, up to 5 years
  collect the data of causes of death and analyze

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Xiao, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Bi N, Ma Y, Xiao J, Zhang H, Xu Y, Tian Y, Li J, Zhang Y, Liu Q, Wang K, Deng L, Wang W, Chen X, Liu F, Zhao R, Yang S, Huang X, Yi J, Hu C, Li Y. A Phase II Trial of Concurrent Temozolomide and Hypofractionated Stereotactic Radiotherapy for Complex Brain Metastases. Oncologist. 2019 Sep;24(9):e914-e920. doi: 10.1634/theoncologist.2018-0702. Epub 2019 Apr 17. PMID 30996008